CLINICAL TRIAL: NCT02902510
Title: Therapeutic Yoga to Improve Function in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00041068
Record Dates: First submitted 2016-09-05; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Parkinson's Disease
Keywords: yoga; function; Parkinson's disease; gait; balance
MeSH Terms: conditions — Parkinson Disease | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): The experimental group is the group that received yoga. The individuals originally assigned to the WLC who completed the yoga intervention AFTER the 8 weeks WLC period also are considered part of the experimental group.
  Interventions: Other: Therapeutic yoga for people with Parkinson's Disease
- Wait List Control (No Intervention): There was no intervention during the WLC.

INTERVENTIONS:
Other: Therapeutic yoga for people with Parkinson's Disease — Held for 8 weeks, individuals participated in therapeutic yoga 60 minutes 2x/week.
  Other Names: Yoga
  Arms: Experimental

SUMMARY:
This is a single blind, randomized, wait-list controlled, phase II exploratory pilot study.

DETAILED DESCRIPTION:
This is a single blind, randomized, wait-list controlled, phase II exploratory pilot study utilizing an after-trial embedded mixed methods approach that will examine the efficacy of therapeutic yoga as a rehabilitation strategy for individuals with PD to improve balance and reduce fear of falling (FoF). Potential participants will have a FoF in order to enter the study. An after-trial embedded mixed methods design will be employed in this study and will include the collection of qualitative data to assist in the overall interpretation of the more heavily weighted quantitative trial data. Adding qualitative methods will serve as a post-hoc analysis capturing participant perceptions of the relationships between the yoga intervention and various outcomes. More specifically, the qualitative data will aide in explaining the link between the various yoga techniques and mechanisms that participants attribute to improved balance, reduced FoF, and other bio-psychosocial outcomes and experiences. Qualitative data will be collected using focus group interviews with participants in the yoga group at the end of the class in week 8.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease with a rating of 1.5-4 on the Modified Hoehn and Yahr Scale of Parkinson's Disease Progression
* Endorsement of FoF,44 able to stand and walk 10 meters with or without an assistive device
* >18 years old; able to speak English
* Score >4 out of 6 on the short Mini Mental Status Exam
* Able and willing to attend twice weekly sessions for 8 weeks

Exclusion Criteria:

* People with self-reported life expectancy <12 months
* Inability to attend sessions due to transportation issues
* Current involvement with other physical activity (including yoga), rehabilitation, or other intervention studies
* Inability or refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Movement Disorders Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  A performance based assessment of motor function.
Change in Mini BESTest at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  clinical balance assessment tool that targets 4 balance control systems, including anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait
Change in Functional Gait Assessment at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  assesses postural stability during 10 walking tasks

SECONDARY OUTCOMES:
Change in Freezing of Gait Questionnaire at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  frequency of freezing of gait and disturbances in gait.
Change in Parkinson's Fatigue Scale at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  measures level of fatigue and impact of fatigue on daily functioning.
Change in Activity Balance Confidence Scale at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  Examines perceived confidence in performing various ambulatory activities with falling.
Change in Activity Constraints Scale at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  Measures perceived constraints to activity participation.
Change in Parkinson's Disease Questionnaire (PDQ-8) at 8 weeks | baseline, 8 weeks (post-intervention), and for individuals in the WLC at the end of the 8-week waiting period
  Measures quality of life for individuals with PD.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Van Puymbroeck, PhD, Principal Investigator — Clemson University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886